CLINICAL TRIAL: NCT01389349
Title: Acupuncture for Tonsillectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's ENT of San Diego, Inc. (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, James W Ochi, M.D., Physician, Children's ENT of San Diego, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2322
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Children; Postoperative Pain; Tonsillar Hypertrophy; Obstructive Sleep Apnea; Chronic Tonsillitis
Keywords: tonsillectomy; adenotonsillectomy; acupuncture; children; postoperative pain; postoperative nausea
MeSH Terms: conditions — Pain, Postoperative; Sleep Apnea, Obstructive; Postoperative Nausea and Vomiting | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Other: Acupuncture
- Sham Control (Sham Comparator)
  Interventions: Other: Sham Control

INTERVENTIONS:
Other: Acupuncture — Battlefield acupuncture protocol
  Arms: Acupuncture
Other: Sham Control — Sham control acupuncture
  Arms: Sham Control

SUMMARY:
Pain after tonsillectomy can be severe and last ten days.

Various new surgical instruments have been developed over the years in an attempt to reduce postoperative pain with mixed results and increased costs; no single tonsillectomy technique is superior to the rest. Patients are discharged to home usually on the day of surgery and often suffer significant pain and nausea. Pain medication is often prescribed which can cause nausea, vomiting and constipation. Children in pain are reluctant to take in fluids and may require intravenous hydration at an emergency department.

"Battlefield acupuncture " has been recently developed by the US Air Force and is now being used in Iraq and Afghanistan on wounded warriors suffering severe acute pain from trauma. This protocol consists of five acupuncture points on the outer ear.

A recent study has demonstrated decreased pain and agitation in children undergoing ear tube insertion. Ear tube patients have mild discomfort compared to tonsillectomy patients and are able to attend school the next day.

The investigators have been encouraged by the benefits of acupuncture during surgery for ear tube patients and also wounded warriors recovering from their injuries. These findings motivated us to see if acupuncture during tonsillectomy surgery would result in less pain and nausea.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 to 17 years of age who need tonsillectomy with or without adenoidectomy with or without myringotomy tube(s)

Exclusion Criteria:

* Developmental Delay

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pain Response | Postoperative days 1 and 6
  Families will be contacted via telephone by a member of the study team other than Dr. Ochi on postoperative days 1 and 6. During these follow-up phone calls a member of the study team will review the daily diary with the parent and also inquire about oral intake, activity level, complications and any additional medical encounters.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Specialty Clinic, El Centro, California
  - Rady Children's Hospital San Diego, San Diego, California